CLINICAL TRIAL: NCT02821832
Title: Using Biomarkers to Predict TB Treatment Duration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 999916133; 16-I-N133
Record Dates: First submitted 2016-06-29; First posted 2016-07-04 (Estimated); Results first posted 2022-12-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Tuberculosis
Keywords: Drug-Resistance; Heteroresistance; Relapse-markers; Medical Imaging; Treatment-shortening
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Urine Specimen Collection; Blood Specimen Collection; Isoniazid; Rifampin; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A - Expected high risk of relapse, standard of care TB treatment (Other): Expected high risk of relapse, standard of care TB treatment
  Interventions: Procedure: Saliva collection; Procedure: Urine collection; Procedure: Sputum collection; Procedure: Blood Collection; Radiation: PET/CT Scan; Drug: Isoniazid, Rifampicin, Pyrazinamide and Ethambutol
- Arm B - Expected low risk of relapse, standard of care TB treatment (Active Comparator): Expected low risk of relapse, standard of care TB treatment
  Interventions: Procedure: Saliva collection; Procedure: Urine collection; Procedure: Sputum collection; Procedure: Blood Collection; Radiation: PET/CT Scan; Drug: Isoniazid, Rifampicin, Pyrazinamide and Ethambutol
- Arm C - Expected low risk of relapse, shortened TB treatment (Experimental): Expected low risk of relapse, shortened TB treatment
  Interventions: Procedure: Saliva collection; Procedure: Urine collection; Procedure: Sputum collection; Procedure: Blood Collection; Radiation: PET/CT Scan; Drug: Isoniazid, Rifampicin, Pyrazinamide and Ethambutol

INTERVENTIONS:
Procedure: Saliva collection — For biomarker assessments
Procedure: Urine collection — For biomarker assessments
Procedure: Sputum collection — For primary endpoint assessments and other biomarker assessments
Procedure: Blood Collection — For biomarker and eligibility assessments
Radiation: PET/CT Scan — Imaging of the lungs to establish disease extent and severity
Drug: Isoniazid, Rifampicin, Pyrazinamide and Ethambutol — Treatment-standard of care

SUMMARY:
Background:

Tuberculosis (TB) is a bacterial lung infection. Typical treatment using anti-TB drugs lasts about 6 months. Some people with less severe TB might not need to take the drugs that long. Researchers think a PET/CT lung scan along with estimating how much TB is in the lungs might show who will be cured after only 4 months of treatment.

Objective:

To demonstrate that 4 months of treatment is not inferior to 6 months of treatment for people with less severe TB.

Eligibility:

People 18-75 years old who have TB treatable with standard TB drugs

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

HIV test

Sputum sample: Participants will be asked to cough sputum into a cup.

Chest x-ray

Participants will start TB drugs. They will have visits at weeks 1, 2, 4, 8, 12, and about 6 more times during the 18-month study. Visits include:

Sputum samples

Physical exam

Blood tests

PET/CT scans at 2-3 visits: Participants fast for about 6 hours before the scan. Participants get FDG, a type of sugar that gives off a small amount of radiation, through an arm vein. They lie on a table in a machine that takes pictures of the body.

Chest x-rays at 1-2 visits

Participants who we believe are likely to be cured at 4 months will be randomly assigned to get either 6 months of treatment or 4 months of treatment.

Participants may be asked to join a substudy using their sputum samples or additional blood tests.

DETAILED DESCRIPTION:
Shortening the duration of treatment for patients with drug sensitive tuberculosis from 6 to 4 months has been attempted many times in clinical trials but thus far all have failed. These failures reveal our incomplete understanding of factors driving the need for such extensive treatments. Consistently, trials have demonstrated that 80-85% of patients are successfully cured after 4 months of therapy, including the extensive set of studies from the British Medical Research Council (BMRC) in the 1970s and 1980, the Tuberculosis Research Unit (TBRU) treatment shortening study in non-cavitary patients who achieve early culture conversion, and the more recent treatment shortening trials using fluoroquinolones like REMoxTB. The current standard of care is to over-treat all patients for a total of 6-months to avoid relapse in a small subset of patients at higher risk for incompletely understood reasons.

For decades, clinical investigators have attempted to establish culture conversion as a predictor of treatment success. Despite the appealing logic, the real correlation of culture conversion as a surrogate endpoint has been consistently disappointing. In the REMoxTB trial, in particular, the intensive microbiological data collected revealed unambiguously that clearance of bacteria from the sputum did not sufficiently correlate with relapse risk to be a useful surrogate for durable cure. An important subset of patients, despite clearing their sputum of TB quickly and complying with all of their medications, still remained at high risk of relapsing with active disease after stopping treatment. Likewise there are patients who clear their sputum of bacteria slowly that nonetheless go on to achieve durable cure. Intuitively this makes sense: only those bacteria at the surface of a cavity are directly open to the airways to seed the sputum. Yet this is not the full story as there are also heterogeneous lesions within each individual patient which respond differently to treatment with chemotherapy.

This protocol builds upon the historical trials and several successful small studies that suggest that directly monitoring lung pathology using (18F)- FDG PET/CT correlates better with treatment outcome than culture status. We will prospectively identify patients at low risk based on their baseline radiographic extent of disease, and further refine this risk score by evaluating the rate of resolution of the lung pathology (CT) and inflammation (PET) at one month as well as checking an end-of-treatment GeneXpert test for the sustained presence of bacteria. Patients classified as low risk will be randomized to receive a shortened 4- month or a full 6-month course of therapy. If successful, this trial will both offer a badly needed alternative to culture status as a trial-level surrogate marker for outcome as well as provide critical information for preclinical and early clinical efforts to identify new agents and combinations with the potential to shorten therapy.

Hypothesis: A combination of radiographic characteristics at baseline, the rate of change of these features at one month, and markers of residual bacterial load at the end of treatment will identify patients with tuberculosis who are cured with 4 months (16 weeks) of standard treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 to 75 years with body weight from 35 kg to 90 kg
  2. Has not been treated for active TB within the past 3 years
  3. Not yet on TB treatment
  4. Xpert positive for M.tb
  5. Rifampin-sensitive pulmonary tuberculosis as indicated by Xpert
  6. Laboratory parameters within previous 14 days before enrollment:

     1. Serum AST and ALT <3x upper limit of normal (ULN)
     2. Creatinine <2x ULN
     3. Hemoglobin >7.0 g/dL
     4. Platelet count >50 x10(9) cells/L
  7. Able and willing to return for follow-up visits
  8. Able and willing to provide informed consent to participate in the study
  9. Willing to undergo an HIV test
  10. At sites with sufficient SARS-CoV-2 testing capacity and personal protective equipment for study staff, willing to undergo COVID-19 testing:

      viral RNA PCR testing for SARS-CoV-2 to determine active infection and antibody testing for SARS-CoV-2 to determine prior infection
  11. Willing to have samples, including DNA, stored
  12. Willing to consistently practice a highly reliable, non-hormonal method of pregnancy prevention (e.g., condoms) during treatment if participant is a premenopausal female unless she has had a hysterectomy or bilateral tubal ligation or her male partner has had a vasectomy. If hormonal contraception is used an additional method of pregnancy prevention (as above) should be used.

EXCLUSION CRITERIA:

1. Clinical suspicion of or confirmed extrapulmonary TB, including pleural TB
2. Pregnant or desiring/trying to become pregnant in the next 6 months or breastfeeding.
3. HIV infected
4. Currently COVID-19 infected
5. Unable to take oral medications
6. Diabetes as defined by point of care HbA1c greater than 6.5%, random glucose greater than 200 mg/dL (or 11.1 mmol/L), fasting plasma glucose greater than or equal to 126 mg/dL (or 7.0 mmol/L), or the presence of any antidiabetic agent (including traditional medicines) as a concomitant medicine
7. Disease complications or concomitant illnesses that may compromise safety or interpretation of trial endpoints, such as known diagnosis of chronic inflammatory condition (e.g. sarcoidosis, rheumatoid arthritis, connective tissue disorder)
8. Use of immunosuppressive medications, such as TNF-alpha inhibitors or systemic or inhaled corticosteroids, within the past 2 weeks
9. Use of any investigational drug in the previous 3 months
10. Substance or alcohol abuse that in the opinion of the investigator may interfere with the participant's adherence to study procedures.
11. Any person for whom the physician feels this study is not appropriate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Clinical Infectious Diseases Research Initiative (Khayelitsha site), Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
.A data sharing committee will be formed to define when and how data will be shared. To protect study integrity, data will not generally be released externally as the study is ongoing, except under extraordinary circumstances. Prior to database lock, data releases will require approval from the data and safety monitoring board, in addition to the data sharing committee. Exceptions to these data release include limited data required for reporting to sponsors (e.g., enrollment updates). After the database has been locked, a formal process for data sharing will be implemented. The data sharing timelines will meet the requirements of the study funders.

REFERENCES:
- [Background] Jindani A, Harrison TS, Nunn AJ, Phillips PP, Churchyard GJ, Charalambous S, Hatherill M, Geldenhuys H, McIlleron HM, Zvada SP, Mungofa S, Shah NA, Zizhou S, Magweta L, Shepherd J, Nyirenda S, van Dijk JH, Clouting HE, Coleman D, Bateson AL, McHugh TD, Butcher PD, Mitchison DA; RIFAQUIN Trial Team. High-dose rifapentine with moxifloxacin for pulmonary tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1599-608. doi: 10.1056/NEJMoa1314210. PMID 25337749
- [Background] Gillespie SH, Crook AM, McHugh TD, Mendel CM, Meredith SK, Murray SR, Pappas F, Phillips PP, Nunn AJ; REMoxTB Consortium. Four-month moxifloxacin-based regimens for drug-sensitive tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1577-87. doi: 10.1056/NEJMoa1407426. Epub 2014 Sep 7. PMID 25196020
- [Background] Merle CS, Fielding K, Sow OB, Gninafon M, Lo MB, Mthiyane T, Odhiambo J, Amukoye E, Bah B, Kassa F, N'Diaye A, Rustomjee R, de Jong BC, Horton J, Perronne C, Sismanidis C, Lapujade O, Olliaro PL, Lienhardt C; OFLOTUB/Gatifloxacin for Tuberculosis Project. A four-month gatifloxacin-containing regimen for treating tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1588-98. doi: 10.1056/NEJMoa1315817. PMID 25337748
- [Derived] Chen RY, Via LE, Dodd LE, Walzl G, Malherbe ST, Loxton AG, Dawson R, Wilkinson RJ, Thienemann F, Tameris M, Hatherill M, Diacon AH, Liu X, Xing J, Jin X, Ma Z, Pan S, Zhang G, Gao Q, Jiang Q, Zhu H, Liang L, Duan H, Song T, Alland D, Tartakovsky M, Rosenthal A, Whalen C, Duvenhage M, Cai Y, Goldfeder LC, Arora K, Smith B, Winter J, Barry Iii CE; Predict TB Study Group. Using biomarkers to predict TB treatment duration (Predict TB): a prospective, randomized, noninferiority, treatment shortening clinical trial. Gates Open Res. 2017 Nov 6;1:9. doi: 10.12688/gatesopenres.12750.1. PMID 29528048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from clinics in and around Cape Town, South Africa (RSA) and Henan Province, China. Recruitment in RSA began on 21Jun2017 and on 17Oct2017 in China. The final participant was recruited for this protocol on 31Mar2021.
Pre-assignment Details: Enrolled participants may have been excluded from participation for the following reasons: identification of baseline drug-resistant TB, withdrawn consent, sputum culture negative on Lowenstein-Jensen medium at baseline, poorly adherent to treatment, developed extrapulmonary TB, or had a significant incidental finding on baseline PET/CT requiring study withdrawal.
Groups:
- Arm A: Expected high risk of relapse based on radiographic criteria, bacterial load criterion, and/or adherence criterion
  standard of care treatment for 6 months: 2 months Isoniazid, Rifampicin, Pyrazinamide and Ethambutol + 4 months Isoniazid, Rifampicin
- Arm B: Expected low risk of relapse based on radiographic criteria, bacterial load criterion, and/or adherence criterion
  standard of care treatment for 6 months: 2 months Isoniazid, Rifampicin, Pyrazinamide and Ethambutol + 4 months Isoniazid, Rifampicin
- Arm C: Expected low risk of relapse based on radiographic criteria, bacterial load criterion, and/or adherence criterion
  shortened treatment: 2 months Isoniazid, Rifampicin, Pyrazinamide and Ethambutol + 2 months Isoniazid, Rifampicin
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 251 | 154 | 141
Completed | 186 | 106 | 109
Not Completed | 65 | 48 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 251 | 154 | 141 | 546
Age, Continuous [Mean (Full Range); unit: years] | 37.5 [18.2 to 75.9] | 35.5 [18.0 to 68.5] | 33.4 [18.4 to 73.8] | 35.8 [18.0 to 75.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 46 | 46 | 150
  Male | 193 | 108 | 95 | 396
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 72 | 55 | 53 | 180
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 179 | 99 | 88 | 366
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 179 | 99 | 88 | 366
  China | 72 | 55 | 53 | 180
Weight [Mean (Standard Deviation); unit: kilograms] | 55.3 (9.5) | 55.0 (9.7) | 57.1 (9.9) | 55.7 (9.7)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 19.5 (2.9) | 19.7 (2.8) | 20.2 (3.2) | 19.7 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Rate of Treatment Success at 18 Months (After Treatment Initiation) Between Arms B and C
Description: Estimation of the lower bound of a one-sided 95% confidence interval of the difference in success rates between arms B and C. If the lower bound is greater than -7%, this will be evidence that the treatment-shortening arm is not inferior to the standard duration arm.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 237 | 132 | 139
Participants
  Cured | 217 | 121 | 117
  Confirmed relapses | 5 | 1 | 9
  Late withdrawal, lost to follow-up | 13 | 9 | 6
  Probable relapses | 1 | 1 | 3
  Treatment Failure | 1 | 0 | 4

2. Secondary Outcome: Radiologic, Immunologic and Microbiologic Measures
Description: The difference (and 95% confidence interval) in treatment success rates between a combined A+B Arm (with Arm A participants selected to represent a true 6-month standard of care population) and a combined Arm A+C (with the remaining Arm A participants selected to represent a treatment shortening strategy arm, and no overlap in Arm A participants assigned to B and C).
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 4/251 | 3/154 | 0/141
Serious Adverse Events (participants affected / at risk) | 20/251 | 5/154 | 3/141
Other Adverse Events (participants affected / at risk) | 0/251 | 0/154 | 0/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=251) | Arm B (N=154) | Arm C (N=141)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gunshot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Head trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic forced the temporary halt of all study activities, which led to some missed visits. As study activities resumed, some study visits and PET/CT scans needed to be done out-of-window. All of the COVID-related protocol deviations can be attributed to clinical site restrictions and safety precautions taken to protect study staff and participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT02821832/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT02821832/SAP_001.pdf